CLINICAL TRIAL: NCT01019200
Title: A Case Control Study to Evaluate Serum Lipid Levels and Other Biomarkers of Cardiovascular Disease in Patients With Psoriasis.
Brief Title: Serum Lipid Levels and Other Biomarkers of Cardiovascular Disease in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#100940
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-02

CONDITIONS: Psoriasis; Cardiovascular Diseases; Dyslipidemia
Keywords: psoriasis; heart disease; cardiovascular disease; hyperlipidemia
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases; Dyslipidemias; Heart Diseases; Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psoriasis: Individuals with a diagnosis of psoriasis as confirmed by the principle investigator will comprise the psoriasis or case group. Participants must meet inclusion and exclusion criteria as defined below. This group will consist of 100 individuals.
- Control: Individuals without psoriasis, but meeting inclusion and exclusion criteria, will be selected to be within the control group. For each patient with psoriasis within the psoriasis group, an age, sex, and BMI-matched control will be selected. The group will consist of 100 individuals.

SUMMARY:
Psoriasis patients are known to be at increased risk for heart disease. This may be due to the increased prevalence of cardiovascular disease risk factors in this population, including high blood pressure, diabetes, obesity, and high cholesterol. Although cholesterol levels are known to be altered in psoriasis, most studies have used standard lipid profiles to measure cholesterol. These tests indirectly measure LDL (bad cholesterol) and become less accurate when triglyceride levels are high, as often see in individuals with psoriasis. We have designed a case-control study that uses a more specific and detailed cholesterol test to measure serum lipid levels in psoriasis patients, allowing for more accurate determination of LDL and better assessment of the lipid-contribution to cardiovascular risk. We will also measure other markers of inflammation that may contribute to cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes from our dermatology clinic, between the age 18 and 80 years who wish to participate voluntarily in the study and who have signed a written informed consent form to participate. Cases will have a diagnosis of psoriasis as diagnosed by our principal investigator, while controls will be selected from the same dermatology clinic.

Exclusion Criteria:

* Current or past use (within 6-8 weeks) of anti-hyperlipidemic agents (statins, fibrates, neomycin, niacin, ezetimibe) and/or any other medications significantly affecting lipid metabolism, including cyclosporine, acitretin, protease inhibitors, tamoxifen, clozapine, and estrogen replacement therapy.
* Presence of secondary causes of hyperlipidemia including diabetes mellitus, smoking, untreated hypothyroidism, nephrotic syndrome, chronic kidney disease, and cholestatic liver disease (e.g. primary biliary cirrhosis).
* History of cardiovascular disease (e.g. previous myocardial infarction, stroke, or angioplasty performed secondary to atherosclerosis).
* History of alcohol intake >30 g/day in males and >20 g/day in females.
* Pregnancy
* Subjects with conditions or diseases hindering data collection and follow up, such as incapacitating diseases, cognitive deterioration, institutionalized patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the Dermatology Clinic at George Washington University Medical Faculty Associates.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2009-11; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Evaluate differences in serum lipid levels in psoriasis patients compared to controls through the use of a relatively new comprehensive lipid profile test that has not been used in previous psoriasis studies. | After consent is obtained

SECONDARY OUTCOMES:
Compare other cardiovascular biomarkers such as high-sensitivity C-Reactive Protein in psoriasis patients verses controls. | After consent is obtained.
Identify if an association exists between the extent and severity of psoriasis and measured lipid levels | After consent is obtained

CONTACTS AND LOCATIONS:
Overall Officials: Alison Ehrlich, MD, Principal Investigator — GWU; Lisa W Martin, MD, Study Chair — GWU; Monica Rengifo-Pardo, Study Chair — GWU
Locations (1):
- The George Washington University Dermatology Clinic, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes